CLINICAL TRIAL: NCT01214356
Title: Impact of Vitamin D on Diabetic Kidney Disease in African Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R03DK089120 (NIH)
Record Dates: First submitted 2010-10-01; First posted 2010-10-05 (Estimated); Results first posted 2018-10-16 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-09

CONDITIONS: Diabetic Kidney Disease
Keywords: diabetes; kidney disease; vitamin D
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus; Kidney Diseases | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Lower Dose Vitamin D (Placebo Comparator): Vitamin D3 supplementation of 400 IU/D or 4000 IU/D with combined calcium carbonate supplementation of 1000 mg/day
  Interventions: Dietary Supplement: Vitamin D3
- Higher Dose Vitamin D (Active Comparator): Vitamin D3 supplementation of 4000 IU/D or 4000 IU/D with combined calcium carbonate supplementation of 1000 mg/day
  Interventions: Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Patients receive vitamin D 400 IU/d with calcium carbonate (1000 mg) once per day for 15 months (3 month run in phase with 12 month follow up)
  Other Names: Cholecalciferol
  Arms: Lower Dose Vitamin D
Dietary Supplement: Vitamin D3 — Patients receive vitamin D 4000 IU/d with calcium carbonate (1000 mg) once per day for 15 months (3 month run in phase with 12 month follow up)
  Other Names: Cholecalciferol
  Arms: Higher Dose Vitamin D

SUMMARY:
This purpose of this project is to evaluate the effectiveness of vitamin D supplementation over 12 months in vitamin D deficient African American adults with type 2 diabetes.

DETAILED DESCRIPTION:
Diabetic kidney disease is increasing in prevalence and is associated with significant morbidity and mortality. Health disparities exist in the progression of diabetic kidney disease, with minorities being more affected even when adjusting for treatment, glycemic and hypertensive control, and medical coverage. Secondary prevention of the progression of diabetic kidney disease is hindered by a lack of easily modifiable risk factors. Based on animal and observational human studies, vitamin D deficiency is potentially a novel, modifiable risk factor that may interrupt or delay the progression of diabetic kidney disease through direct effects as well as by helping to ameliorate kidney disease risk factors, such as hyperglycemia, hypertension and inflammation. In addition, based on minorities having a higher prevalence of vitamin D deficiency, it may also potentially impact the differential progression of diabetic kidney disease in minorities. However, clinical trials evaluating the impact of vitamin D supplementation on diabetic kidney disease are lacking. Thus, this pilot study funded as an R03 through the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) has the following specific aims: (1): To evaluate the impact of vitamin D supplementation (vitamin D3 at 400 IU/d versus 4000 IU/d) on the proportion of individuals with progression of albuminuria over 12 months in a sample of African American participants with vitamin D deficiency in a randomized controlled trial. (2): To identify whether kidney disease risk factors such as blood pressure and glycemic control mediate the impact of vitamin D supplementation on the progression of albuminuria over 12 months in a sample of African American participants with vitamin D deficiency in a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* African American race
* Diagnosis of Type 2 Diabetes
* Stage 1 or 2 Kidney Disease with detectable microalbuminuria >4.0 (mg/g) 25(OH)D level <20 ng/ml

Exclusion Criteria:

* Type 1 diabetes

  --> Stage 3 Kidney Disease, or history of dialysis, kidney transplantation or nephrolithiasis
* Unable to provide informed consent or contact information
* Pre-existing calcium or parathyroid condition, including serum calcium >10.2 mg/dL
* Sarcoidosis, active tuberculosis, or malignancy
* Known hypersensitivity to vitamin D or any of its analogues and derivatives
* Current pregnancy or planning to become pregnant in next 15 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2010-08 (Actual); Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa A Diaz, MD, MS, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible if AA and Vitamin D Deficiency
Pre-assignment Details: eligibility criteria reviewed
Groups:
- Vitamin D: Vitamin D supplementation
- Usual Care: vitamin D3 at 400 IU/d
Period: Overall Study
Arm/Group | Vitamin D | Usual Care
Started | 27 | 27
Completed | 10 | 13
Not Completed | 17 | 14

BASELINE CHARACTERISTICS:
Groups:
- Vitamin D Supplementation: vitamin D3 at 4000 IU/d
- Total: Total of all reporting groups
Arm/Group | Vitamin D Supplementation | Usual Care | Total
Number analyzed (Participants) | 27 | 27 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (10.7) | 53.4 (10.7) | 53.4 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 41
  Male | 7 | 6 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 27 | 27 | 54
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 27 | 27 | 54

OUTCOME MEASURES:

1. Primary Outcome: Change in Urinary Albumin:Creatinine Ratio (ACR)
Description: Urinary Albumin:Creatinine Ratio (ACR) is a well-established, sensitive marker of nephropathy progression (urine albumin (mg/dL) to urine creatinine (g/dL) ratio).
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Vitamin D Supplementation | Usual Care
Number analyzed (Participants) | 10 | 13
ratio | -52.55555556 (151.8477372) | 46.44444444 (47.4125)

2. Secondary Outcome: Decrease in Estimated Glomerular Filtration Rate (eGFR)
Description: Estimated Glomerular Filtration Rate (eGFR) will be evaluated every 6 months, since changes in eGFR and ACR may occur independently and represent different pathways to the development of renal insufficiency. eGFR will be calculated via the Modification of Diet in Renal Disease (MDRD) equation of 4 variables (Cr level, age, sex, race) per NKF recommendations, with serum creatinine (Cr) measured using the SYNCHRON® System by means of the Jaffe rate method. For the purposes of this study, a decrease in eGFR will serve as a secondary outcome measure.
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Vitamin D Supplementation | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/13
Other Adverse Events (participants affected / at risk) | 0/10 | 0/13

LIMITATIONS AND CAVEATS:
small sample size, loss to follow up

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No